CLINICAL TRIAL: NCT04706338
Title: A Study of Transcranial Magnetic Stimulation in the Rehabilitation of Glioma Patients With Postoperative Motor Dysfunction.
Brief Title: Transcranial Magnetic Stimulation in the Rehabilitation of Postoperative Motor Dysfunction.
Acronym: ATM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2020-128-01
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Glioma; Postoperative Motor Deficit
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: patients with postoperative motor deficits, especially for patients with SMA syndrome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TMS treatment (Experimental): Patients with TMS treatment
  Interventions: Device: TMS treatment

INTERVENTIONS:
Device: TMS treatment — Using TMS to stimulate (5 Hz, 90%~110% resting motor threshold) patients' primary motor area and SMA.

SUMMARY:
This study focused on glioma patients with postoperative motor deficits, especially for patients with supplementary motor area syndrome. The investigators want to investigate whether the recovery of motor function will be accelerated by using transcranial magnetic stimulation to stimulate primary motor area and supplementary motor area on the lesional hemisphere.

ELIGIBILITY:
Inclusion Criteria:

1. patient underwent awake craniotomy and motor functional identification during tumor resection;
2. patients with postoperative motor deficit (muscle strength of limbs is weaker than preoperative status)

Exclusion Criteria:

1. patients with contraindication of transcranial magnetic stimulation;
2. patients without data of the pre- and postoperative resting state MRI and diffusion tensor image.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Accelerate motor functional recovery | From the day of tumor resection to 3 months after tumor resection.
  The ratio of motor functional recovery in patients with TMS treatment is higher than those do not receive TMS treatment and the time of motor funcitonal recovery is shorter than those do not receive.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Tao, Study Chair — Beijing Neurosurgical Institute
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The treatment protocal of TMS for glioma patients with postoperative motor dysfunction

REFERENCES:
- [Background] Dionisio A, Duarte IC, Patricio M, Castelo-Branco M. The Use of Repetitive Transcranial Magnetic Stimulation for Stroke Rehabilitation: A Systematic Review. J Stroke Cerebrovasc Dis. 2018 Jan;27(1):1-31. doi: 10.1016/j.jstrokecerebrovasdis.2017.09.008. Epub 2017 Oct 27. PMID 29111342
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449